CLINICAL TRIAL: NCT05783375
Title: Accelerating Delivery of rheUmatic Heart Disease Preventive iNterventions in Northern Uganda
Acronym: ADUNU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Uganda Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-0714
Record Dates: First submitted 2023-02-09; First posted 2023-03-24 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ADUNU Participants (Other): Individuals and healthcare providers residing and working in the involved Ugandan Districts.
  Interventions: Other: ADUNU program for delivery of RHD care services

INTERVENTIONS:
Other: ADUNU program for delivery of RHD care services — The ADUNU program will be deployed by the Ugandan Ministry of Health and the involved District Health Offices to include echocardiography integrated into primary healthcare to screen for RHD and a registry-based care system to keep patients linked to care and prophylaxis.

SUMMARY:
The goal of this prospective study is to evaluate the feasibility, sustainability, and public health impact of a district-based program for secondary prevention of Rheumatic Heart Disease (RHD) in Uganda.

DETAILED DESCRIPTION:
ADUNU is a non-randomized experiment, testing a strategy for implementing an evidence-based practice, decentralized RHD preventive services.

The objectives of the study are to:

Objective 1: Demonstrate the impact of ADUNU, using the RE-AIM framework to assess program Reach, Effectiveness, Adoption, Implementation and Maintenance.

Objective 2: Estimate the cost-effectiveness and budget impact of ADUNU.

ADUNU is a public health initiative that will be deployed the Uganda ministry of health in partnership with the District Health Offices (DHO) in two districts. The program will be overseen by the Technical and Quality Assurance (TAQA). ADUNU's main components will include a RHD testing program which consists of community and facility based echocardiographic screening of children and young adults and a registry based secondary prophylaxis injections of Benzathine penicillin G (BPG) at local health centers III and IVs in both districts.

ELIGIBILITY:
Inclusion Criteria:

* residing in one of two involved districts in Uganda
* providers at HCIIIs and HCIVs located in one of two involved Ugandan districts

Exclusion Criteria:

* None

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 221 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of persons with RHD reached by the ADUNU program | 5 year endpoint
  This objective will involve only secondary analysis of de-identified data collected by districts using routine MOH data collection procedures supplemented by some routine program data during the Ministry's rollout of the ADUNU Programme Package. The number of individuals screened and screening positivity rates will be extracted from screening logs implemented and maintained by DHOs and assessed by modality (school fairs, health days, passive health center screening, and active outreach to family members of RHD diagnosed).
Proportion of persons with RHD enrolled in care, retained and adherent to treatment | 12 months
  Secondary analysis of data from the districts RHD registry will be used to assess the proportion of registrants enrolled, retained and adherent to secondary prophylaxis.
Proportion of persons with RHD enrolled in care, retained and adherent to treatment | 24 months
  Secondary analysis of data from the districts RHD registry will be used to assess the proportion of registrants enrolled, retained and adherent to secondary prophylaxis.
Adoption and implementation of the ADUNU program at the organization level surveys | Baseline
  Brief surveys will be filled out by providers who are acting as administrators of their health centre and will include questions on a range of logistic (e.g., availability of commodities and stockouts, basic infrastructure reliability) and organizational readiness topics (e.g., staffing levels and turnover, organization of patient scheduling, district support visits)
Adoption and implementation of the ADUNU program at the organization level surveys | 24 months
  Brief surveys will be filled out by providers who are acting as administrators of their health centre and will include questions on a range of logistic (e.g., availability of commodities and stockouts, basic infrastructure reliability) and organizational readiness topics (e.g., staffing levels and turnover, organization of patient scheduling, district support visits)
Adoption and implementation of the ADUNU program at the provider level | 6 months
  Two types of data collection activities from frontline providers will be used to understand individual provider-level adoption and maintenance over time: provider surveys and in-depth interviews of providers. A standardized survey instrument on Adoption and a standardized checklist on implementation fidelity that will be completed by the research staff via direct observation. Research staff will use a standardized checklist that will be developed from the core elements of RHD testing (e.g., ultrasound technique, saving of images) and secondary prevention (e.g., injection technique, adequate post-injection monitoring for anaphylaxis)
Adoption and implementation of the ADUNU program at the patient level interview | 24 months
  We will conduct a limited number of interviews of registry patients in each district stratified by adherence outcomes as well as age group (adult vs children).
Cost-analysis of the ADUNU program | 3 year endpoint
  To estimate program costs, we will use the standardized data collection instruments. Our instruments will measure fixed and capital costs, as well as variable or recurrent costs. Ingredients-based costing will be used for drugs and consumables, personnel costs, and equipment costs, whereas gross costing will be used for "indirect" costs such as facility rents and utilities and maintenance. Relevant data for ingredients-based costing include study data on participant healthcare utilization and price lists of drugs, consumables, and equipment. DHO budget sheets for health facilities and overall health service utilization will be used for gross costing. Both financial costs and economic costs will be measured. We will also estimate of out-of-pocket costs borne by registrants, which will allow us to estimate costs from the patient/household perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Z Beaton, Principal Investigator — Cincinnati Chidren's hospital; Emmy H Okello, Principal Investigator — Uganda Heart Institute; David Watkins, Principal Investigator — University of Washington
Locations (1):
- Uganda Heart Institute, Kampala, Uganda, Uganda